CLINICAL TRIAL: NCT03623516
Title: Overdiagnosis of Thyroid Cancer in the Marne and Ardennes Departments of France From 1975 to 2014
Acronym: OTCancer
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao001
Record Dates: First submitted 2018-07-19; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Papillary Thyroid Cancer
Keywords: Thyroid neoplasms; Thyroid gland; ;; Thyroid gland; Incidence; Overdiagnosis
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid cancer: All subjects living in the Marne or Ardennes Departments of France and who were diagnosed with papillary thyroid cancer between 1975 and 2014.

SUMMARY:
Introduction - Incidence of thyroid cancer has increased considerably in France in recent years, but the mortality rate has declined only slightly. Part of this increased incidence could be attributable to overdiagnosis. We aimed to estimate the contribution of overdiagnosis to the incidence of papillary thyroid cancer.

Material and methods. - Incidence rates were calculated based on data from the specialised Marnes-Ardennes thyroid cancer registry, for cancers diagnosed between 1975 and 2014, by age category and by five-year period. The population was divided into two groups according to pTNM classification at diagnosis (i.e. localised or invasive). Overdiagnosis was defined as the difference in incidence rates between the invasive cancer and localised cancer groups. This rate was then divided by the incidence rate in the localised cancer group for the most recent period (2010-2014) to obtain the proportion of cancers attributable to overdiagnosis.

DETAILED DESCRIPTION:
Introduction - Incidence of thyroid cancer has increased considerably in France in recent years, but the mortality rate has declined only slightly. Part of this increased incidence could be attributable to overdiagnosis. We aimed to estimate the contribution of overdiagnosis to the incidence of papillary thyroid cancer.

Material and methods. - We included all subjects living in the Marne or Ardennes Departments of France and who were diagnosed with papillary thyroid cancer between 1975 and 2014. We recorded socio-demographic variables, i.e. age at diagnosis and sex. Cancer characteristics were also recorded, namely year of diagnosis, International Classification of Diseases (ICD) 10th revision code associated with the papillary cancer, and the pTNM 2002 status. Incidence rates were calculated based on data from the specialised Marnes-Ardennes thyroid cancer registry, for cancers diagnosed between 1975 and 2014, by age category and by five-year period. The population was divided into two groups according to pTNM classification at diagnosis (i.e. localised or invasive). Overdiagnosis was defined as the difference in incidence rates between the invasive cancer and localised cancer groups. This rate was then divided by the incidence rate in the localised cancer group for the most recent period (2010-2014) to obtain the proportion of cancers attributable to overdiagnosis.

ELIGIBILITY:
Inclusion Criteria:

* clinical doagnosis of papillary thyroid cancer
* living in the Marne or Ardennes departments of France

Exclusion Criteria:

- cancer stage not determined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects living in the Marne or Ardennes Departments of France and who were diagnosed with papillary thyroid cancer between 1975 and 2014.
Sampling Method: Non-Probability Sample
Enrollment: 2008 (Actual)
Dates: Start 1975-01-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Overdiagnosis of thyroid cancer | 30 years
  Overdiagnosis of thyroid cancer (defined as the diagnosis of disease that would otherwise not go on to cause symptoms or death, and was calculated by comparing the incidence rate of the localised cancer group and that of the invasive cancer group)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Saint-Martin C, Drame M, Dabakuyo S, Kanagaratnam L, Arveux P, Schvartz C. Overdiagnosis of thyroid cancer in the Marne and Ardennes Departments of France from 1975 to 2014. Ann Endocrinol (Paris). 2017 Feb;78(1):27-32. doi: 10.1016/j.ando.2016.07.005. Epub 2016 Sep 15. PMID 27641079